CLINICAL TRIAL: NCT01022827
Title: Effects and Predictors of Effectiveness of Shoulder Muscle Massage for Patients With Posterior Shoulder Stiffness
Brief Title: Shoulder Muscle Massage Shoulder Stiffness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200905041R
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-11

CONDITIONS: Massage Effect
Keywords: stiff shoulder; massage; muscle stiffness
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- posterior shoulder stiffness massage group (Experimental): The inclusion criteria of patients with glenohumeral internal rotation limitation and posterior shoulder stiffness were: [1] limitation of internal rotation ROM compared to the sound side; [2] mild glenohumeral joint hypomobility according to joint play assessment; [3] stiffness in the posterior shoulder region.
  Interventions: Other: massage
- posterior shoulder stiffness placebo group (Placebo Comparator)
  Interventions: Other: massage

INTERVENTIONS:
Other: massage — For the massage group, a physical therapist with 8 years of clinical experience in manual therapy provided the massage on the posterior deltoid, infraspinatus, and teres minor of the involved shoulder for 18 minutes [about 6 minutes for each muscle and order was random] two times a week for 4 weeks. The techniques of massage included petrissage for 3 minutes and rolling for 3 minutes of soft tissues

SUMMARY:
The investigators investigated the effect and predictors of effectiveness of massage in the treatment of patients with posterior shoulder stiffness. This is a randomized controlled trial study- massage and control (hand touch) two times a week for 4 weeks. A total of 60 patients with posterior shoulder tightness were randomized into 2 groups; 52 of them completed this study (29 for the massage and 23 for the control). Patient sex, age, body mass index, glenohumeral internal rotation range of motion (ROM), duration of symptom, functional status, and muscle stiffness were recorded. Additionally, for the massage group, patients with glenohumeral internal rotation improvement of 20 degrees after massage were considered responsive, and the others were considered nonresponsive. The influences of the aftermentioned factors on the effectiveness of massage were analyzed by multivariate logistric regression. The overall mean internal rotation ROM increased significantly after massage (from 31.9° to 54.9°; P < 0.001) compared to the control (from 28.7° to 34.9°; P > 0.05). There were 22 patients in the responsive group and 7 in the nonresponsive group. Among the factors, duration of symptoms, FLEX-SF score, and posterior deltoid stiffness were significant predictors of effectiveness of massage. Massage was an effective treatment for subjects with posterior shoulder stiffness, but was less effective in patients with longer duration of symptoms, higher functional limitation, and less posterior deltoid stiffness.

ELIGIBILITY:
Inclusion Criteria:

1. a limited ROM of internal rotation (internal rotation ROM < 20% to the sound side), and
2. pain and stiffness in the shoulder region for at least 3 months.

Exclusion Criteria:

1. surgery on the particular shoulder,
2. rheumatoid arthritis,
3. stroke with residual shoulder involvement,
4. fracture of the shoulder complex,
5. rotator cuff deficiency, and
6. resting pain, intolerable pain, or muscle spasm during active and/or passive motion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Range of Motion | pre and post-massage

SECONDARY OUTCOMES:
muscle stiffness | pre and post-massage
functional disability | pre and post-massage

CONTACTS AND LOCATIONS:
Overall Officials: JIU-JENQ LIN, PhD, Principal Investigator — School of Physical Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yang JL, Chen SY, Hsieh CL, Lin JJ. Effects and predictors of shoulder muscle massage for patients with posterior shoulder tightness. BMC Musculoskelet Disord. 2012 Mar 27;13:46. doi: 10.1186/1471-2474-13-46. PMID 22449170